CLINICAL TRIAL: NCT03686774
Title: Effect of Oral Administration of Memantine in Pre and Post-surgery in the Prevention of Post-mastectomy Neuropathic Pain
Brief Title: Memantine and Post-mastectomy Neuropathic Pain
Acronym: CLEMANTINE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-407; 2016-004930-75 (Other: 2016-004930-75)
Record Dates: First submitted 2018-09-18; First posted 2018-09-27 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Neuropathic Pain
Keywords: Memantine; post-mastectomy; prophylaxis; Neuropathic pain; Cognitive-emotional parameters
MeSH Terms: conditions — Neuralgia | interventions — Memantine

STUDY DESIGN:
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memantine group (Experimental): Memantine will be given orally for four weeks starting two weeks before surgery. Memantine will be given in increasing doses: 5 mg/day for 3 days; 10 mg/day for 3 days; 15 mg/day for 3 days and 20 mg/day for 5 days.
  Interventions: Drug: Memantine
- Usual care group (Other): Concerning the comparator group, patients will be followed in the same way as those in the "memantine" group except that they will not receive the study treatment.
  Interventions: Other: no memantine

INTERVENTIONS:
Drug: Memantine — Women provide written informed consent prior to their participation in the study, during their Anesthesiology visit. After baseline assessments (15 days before surgery: Day 0 - 15) of pain intensity, cognitive, quality of life and quality of sleep questionnaires, participants will be randomized in two parallel groups: "memantine" (n=75) or "usual care" (n=75). Memantine will be given orally for four weeks starting two weeks before surgery. Endpoints will be assessed 15 days (Day 0 + 15), 3 months (Day 0 + 3 months), 6 months (Day 0 + 6 months) et 12 months (Day 0 + 12 months) post-mastectomy. In order to maintain a good compliance and to verify that women do not develop adverse events, patients will be called once a week by phone. A booklet for monitoring will be completed daily by the patient for 3 months from the day of surgery.
  Arms: Memantine group
Other: no memantine — Concerning the comparator group, patients will be followed in the same way as those in the "memantine" group except that they will not receive the study treatment
  Arms: Usual care group

SUMMARY:
The aim of this study is to evaluate if memantine administered for four weeks starting two weeks before surgery induces a decrease in pain intensity at 3 months post-mastectomy.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label study in patients undergoing mastectomy. Patients included in this trial will receive memantine or not. For patients in the "memantine" group, the treatment will be given in titration (maximum dose of 20 mg/day). Concerning the comparator group, patients will be followed in the same way as those in the "memantine" group except that they will not receive the study treatment. Whether it is the "memantine" group or the "usual care" group, visits will be scheduled under the usual following conditions of the participating center.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years,
* Patient with a diagnosis of breast cancer, programmed for mastectomy with or without axillary dissection and neoadjuvant chemotherapy,
* Patient able to understand and willing to follow the study protocol,
* Acceptance to give a written consent.

Exclusion Criteria:

* Patient with a contraindication to memantine administration (hypertension, severe cardiac or hepatic insufficiency, stroke),
* Patient with diabetes (type I and II),
* Patient with renal insufficiency,
* Patient with drug treatments evaluated by the investigator to be not compatible with the trial,
* Patient treated with specific drugs (amantadine, ketamine, dextromethorphan, L-Dopa, dopaminergic, anticholinergic agonists, barbituric, neuroleptic, IMAO, antispastic agents, dantrolen or baclofen, phenytoin, cimetidine, ranitidine, procainamide, quinidine, quinine, nicotine, hydrochlorothiazide, warfarine),
* Patient with alcohol addiction,
* Epileptic patient or history of epileptic seizure or convulsions,
* Pregnant or nursing woman,
* Patient with a cooperation and an understanding that does not allow for a strict compliance under the conditions set out in the protocol,
* Patient participating in another clinical trial, or being in an exclusion period, or having received a total amount of compensation exceeding 4500 euros over the 12 months preceding the start of the trial,
* Patient benefiting from a legal protection measure (curatorship, guardianship, protection of justice...),

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale (NPRS) | over the 5 days prior to the 3-month post-surgery visit
  The primary endpoint is the measure of the average pain intensity assessed over the 5 days prior to the 3-month post-surgery visit by NPRS, in the "memantine" and "usual care" groups. This scale ranges from 0 no pain to 10 maximal tolerable pain.

SECONDARY OUTCOMES:
Analgesic consumption | Over 12 months
  Post-operative evaluation of analgesic consumption during 12 months, particularly morphine consumption with a daily pain diary and weekly phone call.
Neuropathic pain characteristics | At baseline (15 days before surgery: Day 0 - 15 days), visit 3 (Day 0 + 16 days), visit 4 (Day 0 + 3 months), visit 5 (Day 0 + 6 months) and visit 6 (Day 0 + 12 months).
  Neuropathic Pain in 4 questions" (DN4): DN4 is a clinical tool for the diagnosis of neuropathic pain. This questionnaire has four questions divided into 10 items related to the interview (ie, symptoms) and to the sensory examination (ie, signs). The investigator asks and examines the patient and notes a response "no" or "yes" for each item: "yes" is scored as "1" and "no" is scored as "0". The sum of scores gives the total score of the patient (/10). DN4 is considered as positive if the patient obtains a score of 4/10.
Neuropathic pain evaluation by Neuropathic pain symptom Inventory (NPSI) questionnaire. | At baseline (15 days before surgery: Day 0 - 15 days), visit 3 (Day 0 + 16 days), visit 4 (Day 0 + 3 months), visit 5 (Day 0 + 6 months) and visit 6 (Day 0 + 12 months).
  NPSI is a self-questionnaire and includes 10 pain descriptors. Intensity is rated on 0 to 10 numerical scales and two temporal items are designed to assess spontaneous ongoing pain duration and the number of pain paroxysms over 24 hours. This questionnaire discriminates five distinct clinically relevant dimensions: spontaneous burning pain, spontaneous deep pain, paroxysmal pain, evoked pain, and paresthesia/dysesthesia. Each item is calculated on 10 and the overall test score is scored on 100.
Pain evaluation by the Brief Pain Inventory (BPI). | At baseline (15 days before surgery: Day 0 - 15 days), visit 3 (Day 0 + 16 days), visit 4 (Day 0 + 3 months), visit 5 (Day 0 + 6 months) and visit 6 (Day 0 + 12 months).
  Brief Pain Inventory is a self-administered questionnaire with seven items that measured how much pain interfered with various daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep
Pain evaluation by the McGill Pain questionnaire | At baseline (15 days before surgery: Day 0 - 15 days), visit 3 (Day 0 + 16 days), visit 4 (Day 0 + 3 months), visit 5 (Day 0 + 6 months) and visit 6 (Day 0 + 12 months).
  This questionnaire allows to describe pain experienced during the last 48 hours. It has fifty eight qualifiers divided into sixteen items (A to P). Each qualifier is rated from 0 to 4, where 0 = absent, 1 = low, 2 = moderate, 3 = strong, 4 = very strong. The score is divided between two subclasses, sensory subclass (items A to I) and emotional subclass (items J to P).
Assessment of cognitive parameters by the trail making test (TMT). | At baseline (15 days before surgery: Day 0 - 15 days), visit 3 (Day 0 + 16 days), visit 4 (Day 0 + 3 months), visit 5 (Day 0 + 6 months) and visit 6 (Day 0 + 12 months).
  This non-verbal cognitive test assesses the ability of speed, executive functions, attention, concentration, visual perceptual speed. The test takes place in two parts. In Part A, circles are numbered from 1 to 25 and the patient must connect with lines the numbers in ascending order (1-2-3-4, etc.). In Part B, the circles contain numbers from 1 to 13 and letters from A to L, the patient must connect the circles with lines but alternating numbers and letters (1A-2B -3C, etc.). The patient must connect the circles as quickly as possible for both parts of the test, without lifting the pen from the paper. The TMT B additionally provides an estimate of mental flexibility.
Assessment of cognitive parameters by the Digit symbol substitution test (DSST). | At baseline (15 days before surgery: Day 0 - 15 days), visit 3 (Day 0 + 16 days), visit 4 (Day 0 + 3 months), visit 5 (Day 0 + 6 months) and visit 6 (Day 0 + 12 months).
  DSST is a neuropsychological, nonverbal test, which assesses cognitive deficit and brain damage associated with aging and/or depression. It also evaluates learning ability, concentration and attention. It consists in combining pairs of symbols and numbers as quickly as possible and the score is the correct number of symbols in the time allowed (e.g. 90 or 120 seconds).
Assessment of cognitive parameters with the Functional Assessment of Cancer Therapy Cognitive Function (FACT-COG). | At baseline (15 days before surgery: Day 0 - 15 days), visit 3 (Day 0 + 16 days), visit 4 (Day 0 + 3 months), visit 5 (Day 0 + 6 months) and visit 6 (Day 0 + 12 months).
  The items are rated using a 5-point Likert scale ranged 0 from 4. This questionnaire is composed by four subscales: 2 subscales ranged as following: 0 (never), 1 (one time a week), 2 (two to three times a week), 3 (every day) and 4 (several times a day): Perceived cognitive impairments subscale and comments from others subscale and two others subscale ranged as following: 0 (not at all), 1 (a little), 2 (moderately), 3 (much) and 4 (enormously): Perceived cognitive abilities and impact of quality of life subscales. The total score is obtained with the sum of these 4 subscales
Quality of life assessment by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 items (EORTC QLQ-C30). | At baseline (15 days before surgery: Day 0 - 15 days), visit 3 (Day 0 + 16 days), visit 4 (Day 0 + 3 months), visit 5 (Day 0 + 6 months) and visit 6 (Day 0 + 12 months).
  The average of some questions lead to the score of 15 subscales reported on 100: 9 subscales consisting of several items: 5 subscales measuring functional status (physical, role, social, emotional, cognitive), three subscales measuring symptoms (fatigue, pain, nausea and vomiting) and a global subscale of quality of life and health. Finally, six items/isolated symptoms, covering cancer symptoms and frequent side effects of cancer therapies (e.g. loss of appetite) are also included in the questionnaire. For the 6 item assessing the isolated symptoms and some subscales assessing functional status (as physical, role, social cognitive, emotional) and subscales measuring symptoms (fatigue, pain nausea and vomiting): higher values represent a worse outcome. Concerning subscale of quality of life and health, higher values represent a better outcome.
Anxiety and depression assessment with the Hospital Anxiety and Depression scale (HAD). | At baseline (15 days before surgery: Day 0 - 15 days), visit 3 (Day 0 + 16 days), visit 4 (Day 0 + 3 months), visit 5 (Day 0 + 6 months) and visit 6 (Day 0 + 12 months).
  The anxiety sub-score is obtained by summing items relate to anxiety (Subscore Anxiety (A): /21). The depression sub-score is obtained by summing items relate to depression (subscore Depression: /21). For each of the two subscores, if a subject obtain a score ranged from: 0 to 7, he is considered as "normal"; 8-10 = Borderline abnormal (borderline case) and 11-21 = Abnormal (case).
Sleep assessment with the Pittsburgh Sleep Quality Index (PSQI) | At baseline (15 days before surgery: Day 0 - 15 days), visit 3 (Day 0 + 16 days), visit 4 (Day 0 + 3 months), visit 5 (Day 0 + 6 months) and visit 6 (Day 0 + 12 months).
  The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication and daytime dysfunction).In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France